CLINICAL TRIAL: NCT05550935
Title: Effects of High-flow Nasal Cannula on the Distribution of Pulmonary Ventilation and Respiratory Effort in Healthy Subjects During Exercise.
Brief Title: Physiological Effects of High-flow Nasal Cannula During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 220510003
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: High-Flow Nasal Cannula; Electrical Impedance Tomography; Respiratory Physiology; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants receive one of two alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study
Masking Description: An attempt will be made to keep the research team performing the measurements masked to the healthy subject assignment until the first day of the Constant Work-Rate Exercise Test (first random order).
  An attempt will be made to keep the participant masked by simulation with HFNC at 2 L/min and separation of one week between the two exercise tests to forget the effect of the high flow and sound of the device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC Group (Experimental): Healthy subject will perform one Constant Work-Rate Exercise Test at respiratory compensation point as determined by a cardiopulmonary exercise test with High Flow Nasal at 60L/min (without additional oxygen)
  Interventions: Device: High-flow Nasal Cannula
- Control Group (Sham Comparator): Healthy subject will perform one Constant Work-Rate Exercise Test at respiratory compensation point as determined by a cardiopulmonary exercise test with High Flow Nasal at 2L/min (without additional oxygen)
  Interventions: Device: High-flow Nasal Cannula

INTERVENTIONS:
Device: High-flow Nasal Cannula — HFNC is a device that, in this study, will give the maximum flow (60 L/min), with minimum adjusted temperature (31°C) and FiO2 of 21% or room air.
  Other Names: HFNC

SUMMARY:
The high-flow nasal cannula (HFNC) has increased its evidence in patients during pulmonary rehabilitation. These studies hypothesize that the physiological effects of HFNC (positive expiratory pressure, anatomical dead space lavage, thermo-humidification) lead to an increase in exercise time. This is believed to be due to improvements that the device can generate in the respiratory system and muscles. However, the physiological effects of HFNC on respiratory effort and distribution of pulmonary ventilation during exercise are unknown. The aim of this study is to determine the acute effect of high flow nasal cannula on the distribution of pulmonary ventilation and respiratory effort during physical exercise in healthy subjects.

DETAILED DESCRIPTION:
A randomized, cross-over clinical trial in which either HFNC or Sham may be used as an adjunct on a cycle ergometer in random order will be performed to compare the respiratory effort and distribution of pulmonary ventilation continuously. Measurements will be taken in a warm-up, exercise, and recovery phase for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults volunteers
* Physically inactive (according to World Health Organization criteria).

Exclusion Criteria:

* Refusal to participate
* Smokers
* History of acute cardiorespiratory or musculoskeletal disease during the last year (including COVID-19 when hospitalization or supplemental oxygen was required without any other disease)
* Any neuromuscular or cardiovascular or condition that limits test performance.
* Contraindication for esophageal catheter installation (recent epistaxis, severe coagulopathy, among other).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
Inspiratory effort | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  The average esophageal pressure swings during inspiration (ΔPes) defined as the absolute differences between end-expiratory and end-inspiratory Pes over a period of 60 seconds. Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Standard deviation of regional ventilation delay index (RVDsd) | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  as a measure of temporal distribution of ventilation: defined as the average of 10 breaths representative of the 60 seconds evaluated in each period. Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.

SECONDARY OUTCOMES:
Work of breathing | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  The average pressure time product over a minute (PTPmin), defined as the sum of the areas subtended by the Pes waveform during inspiration over 60 seconds. Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Work of breathing per single breath | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  The average per-breath pressure time product (PTP), defined as the area subtended by the Pes waveform during inspiration in a series of representative and valid breaths divided by the number of breaths (at least five to ten) over 60 seconds. Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Respiratory drive | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  The average of negative pressure measured 500 ms after the initiation of an inspiratory effort defined as the defection in Pes during the first 0.5 s during inspiration in a series of representative and valid breaths divided by the number of breaths (at least five to ten) over 60 seconds. Also, The average slope of the inspiratory negative Pes swings from the start of inspiration to the minimum pressure (ΔPes/Δt) in a series of representative and valid breaths divided by the number of breaths (at least five to ten) over 60 seconds.
  Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Tidal Variation (TV) as a measure of variation during tidal breathing | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  defined as the average of differences between end-expiratory lung impedance (EELI) and end-inspiratory lung impedance (EILV) in 60 seconds for each period evaluated warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
End-Expiratory Lung Impedance (EELI), as a measure lung aeration | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  average of end-expiratory lung impedance respectively, in 60 seconds for each period evaluated warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Normalized Tidal Variation (TV) as a measure of variation during tidal breathing | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  defined as the average of differences between end-expiratory lung impedance (EELI) and end-inspiratory lung impedance (EILV) divided by the number of breaths evaluated in each period (60 seconds).Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Normalized End-Expiratory Lung Impedance (EELI) | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  as a measure lung aeration: defined as the average of end-expiratory lung impedance divided by the number of breaths evaluated in each period (60 seconds). Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Global inhomogeneity index (GI) as a measure of spatial distribution of tidal ventilation | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  defined as the value of the tidal image in 60 seconds for each period evaluated. Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Center of ventilation (COV), dorsal fraction of ventilation (TVd) and anterior-to-posterior ventilation ratio (Impedance ratio), most dorsal region of interest (ROI4) (TVroi4), as a measure of ventilation distribution influenced by gravity. | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  defined as the value of the tidal image in 60 seconds for each period evaluated. Measurements will be during warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Dyspnea and leg fatigue | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  : using Modified Borg Scale (0 - 10 points) for each period evaluated warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Heart rate | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  using a pulse oximetry for each period evaluated warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Pulse oxygen saturation | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  using a pulse oximetry for each period evaluated warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Respiratory rate | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during warm-up, exercise, and recovery
  using a electrical impedance tomography for each period evaluated warm-up (one minute of five minutes), exercise (minutes: 0-1'; 3-4'; 5-6'), and the recovery phase (minutes: 0-1'; 1-2'; 3-4'; 5-6';7-8';9-10') for both groups.
Blood pressure | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately seven days, for a total time frame of 3 weeks maximum per participant. Data will be collected during the basal and recovery phase
  Using a sphygmomanometer and stethoscope will be evaluated at the beginning (basal), end of the exercise, and during the recovery phase by the same operator.
Comfort scale associated with dispositive | at 3 weeks. Outcome will be measured during the CWRET and will be carried out on different days, separate from approximately 7 days, for a total time frame of 3 weeks maximum per participant. Data will be collected during the basal and end-exercise
  using visual analog likert scale (0-5: 0: "nothing comfortable" to 5: "totally comfortable") evaluated before and at the end of the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Garcia, PhD(C), Principal Investigator — Departamento Ciencias de la Salud, Facultad de Medicina, Pontificia Universidad Católica de Chile.
Locations (1):
- Laboratorio de Fisiología del Ejercicio, Departamento Ciencias de la Salud, Facultad de Medicina, Pontificia Universidad Católica de Chile., Santiago, Provincia, Chile

IPD SHARING:
Plan to Share IPD: No
The investigators will evaluate IPD sharing since it is not intended a priori to perform an inferential analysis with statistics to evaluate the results before completing the study. In addition, it is a physiological study requiring only three days per subject (Approximately three weeks total) and with a low sample size.